CLINICAL TRIAL: NCT04210895
Title: Efficacy of Footbaths With Ginger Powder on Subjectively Perceived Quality of Sleep: a Randomized Controlled Pilot Study
Brief Title: Efficacy of Footbaths With Ginger Powder on Subjectively Perceived Quality of Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INS_01
Record Dates: First submitted 2019-12-18; First posted 2019-12-26 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Nonorganic Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm footbath with ginger powder (Experimental): Participants receive a daily warm water footbath with added ginger powder over a two-week period
  Interventions: Other: Ginger powder footbath
- Warm water only footbath (Active Comparator): Participants receive a daily warm water footbath over a two-week period
  Interventions: Other: Warm water only footbath

INTERVENTIONS:
Other: Ginger powder footbath — 40 ± 2 ° C warm water footbath with an additive of dried ginger powder reaching up to mid-calf level
  Arms: Warm footbath with ginger powder
Other: Warm water only footbath — 40 ± 2 ° C warm water footbath without any additive reaching up to mid-calf level
  Arms: Warm water only footbath

SUMMARY:
A randomized, controlled trial to explore whether warm footbaths with added ginger powder can improve the sleep quality of adults with self-perceived insomnia symptoms. Participants receive daily footbaths either with warm water alone or with added ginger powder over a period of 2 weeks.

DETAILED DESCRIPTION:
This is a randomized controlled trial with parallel group design to explore the effects of warm water footbaths with added ginger powder (experimental) compared to footbaths with warm water alone (active comparator) on sleep quality in adults with self-perceived insomnia symptoms. Participants receive daily footbaths 1-3 hours before bedtime over a period of two weeks. The footbaths are prepared by the participants themselves and carried out at their homes. Outcome measures are assessed at baseline (pre intervention) and two weeks after baseline (post intervention). The main focus is on change in subjective quality of sleep as assessed by the Pittsburgh Sleep Quality Index (PSQI). The statistical analysis comprises analyses of variance based on linear mixed effects models.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* age between 18 and 70 years
* self-reported insomnia symptoms

Exclusion Criteria:

* known organic insomnia (e.g. periodic leg movements during sleep, restless legs syndrome, sleep apnea syndrome, narcolepsy)
* current intake of allopathic hypnotics
* shift work
* skin lesions at the lower legs or feet
* known intolerance or hypersensitivity to ginger preparations
* acute mental disorder
* varicose vein (degree 3 or 4, classification according to Marshall), chronic venous insufficiency
* pregnancy
* participation in other studies
* insufficient knowledge of the german language

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-04-11 (Actual); Study Completion 2020-04-11 (Actual)

PRIMARY OUTCOMES:
Change in global PSQI Score | Baseline (pre intervention), 2 weeks after baseline (post intervention)
  Global score of the Pittsburgh Sleep Quality Index, score between 0=positive extreme and 21=negative extreme

SECONDARY OUTCOMES:
Change in subjective sleep quality as assessed by the Pittsburgh Sleep Quality Index (PSQI) | Baseline (pre intervention), 2 weeks after baseline (post intervention)
  Scale of the Pittsburgh Sleep Quality Index, score between 0=positive extreme and 3=negative extreme
Change in sleep latency as assessed by the PSQI | Baseline (pre intervention), 2 weeks after baseline (post intervention)
  Scale of the Pittsburgh Sleep Quality Index, score between 0=positive extreme and 3=negative extreme
Change in sleep duration as assessed by the PSQI | Baseline (pre intervention), 2 weeks after baseline (post intervention)
  Scale of the Pittsburgh Sleep Quality Index, score between 0=positive extreme and 3=negative extreme
Change in sleep efficiency as assessed by the PSQI | Baseline (pre intervention), 2 weeks after baseline (post intervention)
  Scale of the Pittsburgh Sleep Quality Index, score between 0=positive extreme and 3=negative extreme
Change in sleep disturbance as assessed by the PSQI | Baseline (pre intervention), 2 weeks after baseline (post intervention)
  Scale of the Pittsburgh Sleep Quality Index, score between 0=positive extreme and 3=negative extreme
Change in use of sleep medication as assessed by the PSQI | Baseline (pre intervention), 2 weeks after baseline (post intervention)
  Scale of the Pittsburgh Sleep Quality Index, score between 0=positive extreme and 3=negative extreme
Change in daytime dysfunction as assessed by the PSQI | Baseline (pre intervention), 2 weeks after baseline (post intervention)
  Scale of the Pittsburgh Sleep Quality Index, score between 0=positive extreme and 3=negative extreme
Change in the Insomnia Severity Index total score | Baseline (pre intervention), 2 weeks after baseline (post intervention)
  Total score of the Insomnia Severity Index, score between 0=no clinically significant insomnia and 28=severe clinical insomnia
Evening protocol: Change in general well-being as assessed by a standardized sleep diary | In the evening (before going to sleep), during the two-week intervention phase between pre intervention (baseline) and post intervention (2 weeks after baseline)
  Self-reported well-being measured with a standardized sleep diary (six-point rating scale, higher values represent a better outcome)
Evening protocol: Change in the average performance as assessed by a standardized sleep diary | In the evening (before going to sleep), during the two-week intervention phase between pre intervention (baseline) and post intervention (2 weeks after baseline)
  Self-reported performance measured with a standardized sleep diary (six-point rating scale, lower values represent a better outcome)
Evening protocol: Change in fatigue as assessed by a standardized sleep diary | In the evening (before going to sleep), during the two-week intervention phase between pre intervention (baseline) and post intervention (2 weeks after baseline)
  Self-reported fatigue measured with a standardized sleep diary (four-point rating scale, lower values represent a better outcome)
Evening protocol: Change in sleep during daytime as assessed by a standardized sleep diary | In the evening (before going to sleep), during the two-week intervention phase between pre intervention (baseline) and post intervention (2 weeks after baseline)
  Self-reported sleep during daytime measured with a standardized sleep diary (specification in minutes, lower values represent a better outcome)
Morning protocol: Change in recovery ability as assessed by a standardized sleep diary | In the morning (after waking up), during the two-week intervention phase between pre intervention (baseline) and post intervention (2 weeks after baseline)
  Self-reported recovery ability measured with a standardized sleep diary (five-point rating scale, lower values represent a better outcome)
Morning protocol: Change in general well-being as assessed by a standardized sleep diary | In the morning (after waking up), during the two-week intervention phase between pre intervention (baseline) and post intervention (2 weeks after baseline)
  Self-reported well-being measured with a standardized sleep diary (six-point rating scale, higher values represent a better outcome)
Morning protocol: Change in sleep latency as assessed by a standardized sleep diary | In the morning (after waking up), during the two-week intervention phase between pre intervention (baseline) and post intervention (2 weeks after baseline)
  Self-reported sleep latency measured with a standardized sleep diary (specification in minutes, lower values represent a better outcome)
Morning protocol: Change in nocturnal awakening as assessed by a standardized sleep diary | In the morning (after waking up), during the two-week intervention phase between pre intervention (baseline) and post intervention (2 weeks after baseline)
  Self-reported nocturnal awakening measured with a standardized sleep diary (specification in minutes, lower values represent a better outcome)
Morning protocol: Change in sleep duration as assessed by a standardized sleep diary | In the morning (after waking up), during the two-week intervention phase between pre intervention (baseline) and post intervention (2 weeks after baseline)
  Self-reported sleep duration measured with a standardized sleep diary (specification in hours, higher values represent a better outcome)
Change in quality of life as assessed by the 12-Item Short Form Survey | Baseline (pre intervention), 2 weeks after baseline (post intervention)
  Scales of the 12-Item Short Form Survey (SF-12), scores between 0=more dysfunction/impairment and 100=less dysfunction/impairment
Change in subjective feeling of overall warmth as assessed by the Herdecke Warmth Perception Questionnaire | Baseline (pre intervention), 2 weeks after baseline (post intervention)
  Self-reported feeling of overall warmth and warmth at the face, trunk anterior/posterior, hands and feet measured with the Herdecke Warmth Perception Questionnaire, scores between 0=cold and 4=hot
Heart rate variability analysis (HRV): Change in RMSSD | Baseline (pre intervention) and two weeks after baseline (post intervention)
  Root mean square of successive differences (RMSSD) [ms]. HRV data are obtained from 24-hour ECG measurements with "Cardioscout Multi-ECG" (SR-Medizinelektronik, Stuttgart, Germany)
Heart rate variability analysis (HRV): Change in SDNN | Baseline (pre intervention) and two weeks after baseline (post intervention)
  Standard deviation of normal to normal (NN) intervals (SDNN) [ms]. HRV data are obtained from 24-hour ECG measurements with "Cardioscout Multi-ECG" (SR-Medizinelektronik, Stuttgart, Germany)
Heart rate variability analysis (HRV): Change in pNN50 | Baseline (pre intervention) and two weeks after baseline (post intervention)
  The proportion of NN50 (number of pairs of successive NNs that differ by more than 50 ms) divided by total number of NNs (pNN50). HRV data are obtained from 24-hour ECG measurements with "Cardioscout Multi-ECG" (SR-Medizinelektronik, Stuttgart, Germany)
Heart rate variability analysis (HRV): Change in VLF | Baseline (pre intervention) and two weeks after baseline (post intervention)
  Very low frequency (VLF, 0.0033 to 0.04 Hz) from frequency domain analysis. HRV data are obtained from 24-hour ECG measurements with "Cardioscout Multi-ECG" (SR-Medizinelektronik, Stuttgart, Germany)
Heart rate variability analysis (HRV): Change in LF | Baseline (pre intervention) and two weeks after baseline (post intervention)
  Low frequency (LF, 0.04 to 0.15 Hz) from frequency domain analysis. HRV data are obtained from 24-hour ECG measurements with "Cardioscout Multi-ECG" (SR-Medizinelektronik, Stuttgart, Germany)
Heart rate variability analysis (HRV): Change in HF | Baseline (pre intervention) and two weeks after baseline (post intervention)
  High frequency (HF, 0.15 to 0.40 Hz) from frequency domain analysis. HRV data are obtained from 24-hour ECG measurements with "Cardioscout Multi-ECG" (SR-Medizinelektronik, Stuttgart, Germany)
Heart rate variability analysis (HRV): Change in LF/HF ratio | Baseline (pre intervention) and two weeks after baseline (post intervention)
  Ratio of two bands from frequency domain analysis: LF band (0.04 to 0.15 Hz) and HF band (0.15 to 0.40 Hz). HRV data are obtained from 24-hour ECG measurements with "Cardioscout Multi-ECG" (SR-Medizinelektronik, Stuttgart, Germany)
Change in distal-proximal skin-temperature gradient | Baseline (pre intervention) and two weeks after baseline (post intervention)
  24-hour measurement of the skin temperature at the feet and abdomen with "MAXIM I-Button™ DS1922L" (Maxim integrated, San Jose, USA). The gradient is calculated by subtracting the proximal value from the distal value.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vagedes, MD, Study Director — ARCIM Institute
Locations (1):
- Arcim Institute, Filderstadt, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be made available, in addition to study protocol and informed consent form.
Supporting Information: Study Protocol, ICF
Time Frame: The data will be made available upon publication for a duration of three months.
Access Criteria: The data will be made available to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal.